CLINICAL TRIAL: NCT02217839
Title: Multiple Ascending Dose Tolerability, Pharmacokinetic and Pharmacodynamic Study of DG3173
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aspireo Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DG3173-I-002
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — PTR 3173; Octreotide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DG3173 (Experimental)
  Interventions: Drug: DG3173; Drug: Octreotide; Drug: DG3173 Placebo
- DG3173+Octreotide (Experimental)
  Interventions: Drug: DG3173+Octreotide; Drug: DG3173 Placebo+Octreotide Placebo; Drug: Octreotide+DG3173 Placebo

INTERVENTIONS:
Drug: DG3173
  Arms: DG3173
Drug: DG3173+Octreotide
  Arms: DG3173+Octreotide
Drug: Octreotide
  Arms: DG3173
Drug: DG3173 Placebo
  Arms: DG3173
Drug: DG3173 Placebo+Octreotide Placebo
  Arms: DG3173+Octreotide
Drug: Octreotide+DG3173 Placebo
  Arms: DG3173+Octreotide

SUMMARY:
This multi-ascending dose study is designed to investigate the safety, tolerability, pharmacokinetic and side effect profile of multiple ascending doses of DG3173, in up to 48 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic origin: Caucasian
* Body Mass Index (BMI): 19-27 kg/m2 inclusive
* Medical history without clinically relevant pathologies
* Physical examination parameters without signs of clinically relevant pathologies
* Electrocardiogram recording without signs of clinically relevant pathology, in particular QTc (Bazett) <450 ms
* Values for hematology and for biochemistry tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator (in particular for alanine transaminase, aspartate transaminase, lactate dehydrogenase, gamma glutamyl transferase, alkaline phosphatase, bilirubin, and α-amylase)
* Subjects with partner of child bearing potential must be willing to practice a medically approved method of contraception (e.g., condom in combination with hormonal contraception or intrauterine device or a diaphragm with spermicide after the first drug administration and for one month after participation in the study or are vasectomized since > 6 months or has a partner being sterilized since > 6 months
* Having given written informed consent before any study related activities are carried out

Exclusion Criteria:

* Evidence of clinically relevant pathology or disease
* Any history of moderate or severe hypertension, hypotension or orthostatic hypotension
* Mental handicap
* Legal incapacity
* Any history of clinically important emotional and/or psychiatric illness or of any clinically important neurological disorders and/or epilepsy
* Chronic diarrhea or other acute or chronic gastrointestinal disorders
* Presence or history of endocrine disorders
* Presence or history of gallstone disease
* Known hypersensitivity to the study drug or constituent of the study drug
* History of any relevant allergy, especially drug and/or food allergies
* Strict vegetarian
* Regular treatment with medications during three months prior to randomization
* Receipt of any prescription or non-prescription medication, including multi vitamin preparations within 14 days prior randomization and for the duration of the study
* Use of St. John's Wort or Ginkgo Biloba (also known as Ginkgo Bilbao) within 48 hours prior to randomization
* Participation in a clinical study within 30 days prior to randomization
* Donation of blood within 60 days prior to randomization
* Receipt of blood, blood products or plasma derivates one year prior to randomization
* Regular smoking of >5 cigarettes per day within the past three months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events or withdrawals due to adverse events. Laboratory investigations (including biochemistry, hematology, and urinalysis), vital signs (blood pressure, pulse rate), and 12-lead ECG. | 10 days